CLINICAL TRIAL: NCT04638075
Title: Use of Supplemental Nursing System Compared to Bottle Supplementation on Breastfeeding Rates in Hospitalized Neonates With Hyperbilirubinemia
Brief Title: Supplemental Nursing System Compared to Bottle Supplementation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to COVID-19 public health crisis.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-0185
Record Dates: First submitted 2020-09-28; First posted 2020-11-20 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Breast Feeding, Exclusive
Keywords: Supplemental Nursing System
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial comparing the SNS to bottle feeding. Once eligibility is determined and consent is obtained, the Primary Investigator (PI)/ Co-Investigator (CI) will randomize the mother-neonate dyad to either bottle supplemental feedings (group A) or SNS supplemental feedings (group B). Randomization will be done by using a computer-generated table of random numbers. Breast milk feeding and exclusive breastfeeding rates will be compared between both groups during the last 24 hours of hospitalization, at day of life 14 and at day of life 28.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A Bottle Supplementation (No Intervention): Group A will supplement using the bottle. The mother will breastfeed as frequently as the neonate's physician allows. When the physician recommends supplementation, the mother will supplement using the bottle per standard of care. The mother will breastfeed for up to 25 minutes and then will offer a bottle to supplement breastfeeding for at least 5 minutes. Time at the breast and with the bottle might vary based on the neonate's ability to stay awake at the breast and to sustain a latch at the breast. The type of supplementation will be either Expressed Breast Milk (EBM), Donor Human Milk (DHM), formula, or a combination of EBM and formula or EBM and DHM. The volume of supplementation and duration of bottle use will be determined by the neonate's physician. The mother will return the neonate to their crib then pump and hand express after feeding sessions per the IBCLC's recommendation. The mother will document each feeding session in the feeding log provided at the bedside.
- Group B SNS Supplementation (Experimental): Group B will supplement using the SNS. The mother will breastfeed as frequently as the neonate's physician allows. When the physician recommends supplementation, the mother will supplement using the SNS per standard of care. The mother will assemble the SNS, place it clamped and in position at the nipple prior to breastfeeding (see SNS instructions for use). The mother will initiate breastfeeding for up to 5 minutes and then unclamp the SNS to begin supplementation for up to 25 minutes. The SNS will contain either EBM, DHM, formula, or a combination of EBM and formula or EBM and DHM. The volume of supplementation and duration of SNS use will be determined by the neonate's physician. The mother will pump and hand express after feeding sessions per the IBCLC's recommendation. Them mother will document each feeding session in the feeding log provided at the bedside.
  Interventions: Device: Supplemental Nursing System

INTERVENTIONS:
Device: Supplemental Nursing System — The SNS is a device designed to deliver supplemental milk by suckling at the mother's nipple. A specially designed bottle attaches to the mother's breast and serves as the reservoir for milk. Attached to the bottle is a small tube which runs down to and is placed on the tip of the mother's nipple. With an adequate latch the neonate obtains supplementation by suckling. Additionally, this suckling stimulates milk production (Lawrence & Lawrence, 2016).
  Arms: Group B SNS Supplementation

SUMMARY:
This is a randomized controlled trial comparing the SNS to bottle feeding. This study will compare exclusive breastfeeding rates and breast milk feeding rates at discharge, day of life 14, and day of life 28 between neonates hospitalized in the NICU for hyperbilirubinemia between those who receive supplementation by the (SNS) or those who receive supplementation by bottle. Additionally, this study will evaluate mothers' experiences while using the SNS. We hypothesize mothers who utilize the SNS will have higher rates of breast milk feeding compared to mothers who supplement by bottle.

DETAILED DESCRIPTION:
Supplemental feedings in the neonatal intensive care unit (NICU) are common due to the separation of mother and neonate and/or complex medical issues that make direct breastfeeding difficult. The Supplemental Nursing System (SNS) is utilized infrequently in the NICU and there is little data available to compare breastfeeding outcomes of mothers who supplement by bottle compared to SNS. The aims of this study are to understand whether supplementation by SNS improves breastfeeding outcomes compared to neonates supplemented by bottle. From December 1, 2018 - November 30, 2019 there were 195 neonates admitted to Children's Hospital Colorado (CHCO) with a primary diagnosis of hyperbilirubinemia who were born at 37 weeks or greater. This makes up approximately 13.7% of all admissions during that time frame. This is a population of mothers at risk for cessation of exclusive breastfeeding due to the necessity of supplementation. These neonates are frequently supplemented because the mother's milk typically is not yet in to support adequate nutritional intake. These neonates are not often medically complex or have any factors that would bias the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* Neonate inclusion criteria: physician diagnosis of hyperbilirubinemia, otherwise healthy term neonates (gestational age 38 weeks +), appropriate size for gestation, and good latch to mother's nipple, with some consistent suckling behavior per standard assessment.

Maternal inclusion criteria: English or Spanish Speaking (with the use of medical interpreter), 18 years of age or greater, desire to exclusively breast milk feed, and must be available at the bedside for all feeding sessions during hospitalization.

Exclusion Criteria:

* Neonate exclusion criteria: Breast milk jaundice, and any condition that prevents the neonate from breastfeeding efficiently including anatomical abnormalities (cleft lip, cleft palate), neurological impairment, symptomatic hypoglycemia, newly diagnosed infections, cardiac anomalies, and intravenous fluid hydration.

Maternal exclusion criteria: Retained placenta, history of breast reduction surgery or breast radiation, physician diagnosed Sheehan's Syndrome, known hypoplastic breast tissue with a low supply after previous deliveries.

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Breastfeeding During Hospitalization | The Daily Feeding Log measures breastfeeding rates from within 12 hours after hospital admission to discharge, an average of 3 days.
  The Daily Feeding Log measures the frequency and duration of breastfeeding.
Rate of Exclusive Breastfeeding at Day of Life 14. | The rate of exclusive breastfeeding is measured from hospital discharge to day of life 14.
  A survey is sent out at day of life 14 with a yes/no maternal response to a question asking if mother is exclusively breastfeeding.
Rate of Exclusive Breastfeeding at Day of Life 28. | The rate of exclusive breastfeeding is measured from day of life 14 to day of life 28.
  A survey is sent out at day of life 28 with a yes/no maternal response to a question asking if mother is exclusively breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bonavita, BSN, Principal Investigator — Colorado University

IPD SHARING:
Plan to Share IPD: No
This data will be maintained at Children's Hospital Colorado only at this time.

REFERENCES:
- [Background] Bar S, Milanaik R, Adesman A. Long-term neurodevelopmental benefits of breastfeeding. Curr Opin Pediatr. 2016 Aug;28(4):559-66. doi: 10.1097/MOP.0000000000000389. PMID 27386975
- [Background] Bertini G, Dani C, Tronchin M, Rubaltelli FF. Is breastfeeding really favoring early neonatal jaundice? Pediatrics. 2001 Mar;107(3):E41. doi: 10.1542/peds.107.3.e41. PMID 11230622
- [Background] Binns C, Lee M, Low WY. The Long-Term Public Health Benefits of Breastfeeding. Asia Pac J Public Health. 2016 Jan;28(1):7-14. doi: 10.1177/1010539515624964. PMID 26792873
- [Background] Borucki LC. Breastfeeding mothers' experiences using a supplemental feeding tube device: finding an alternative. J Hum Lact. 2005 Nov;21(4):429-38. doi: 10.1177/0890334405277822. PMID 16280559
- [Background] Chaturvedi P. Relactation. Indian Pediatr. 1994 Jul;31(7):858-60. PMID 7890356
- [Background] Cheales-Siebenaler NJ. Induced lactation in an adoptive mother. J Hum Lact. 1999 Mar;15(1):41-3. doi: 10.1177/089033449901500111. PMID 10578774
- [Background] Flaherman VJ, Maisels MJ; Academy of Breastfeeding Medicine. ABM Clinical Protocol #22: Guidelines for Management of Jaundice in the Breastfeeding Infant 35 Weeks or More of Gestation-Revised 2017. Breastfeed Med. 2017 Jun;12(5):250-257. doi: 10.1089/bfm.2017.29042.vjf. Epub 2017 Apr 10. No abstract available. PMID 29624434
- [Background] Howard CR, Howard FM, Lanphear B, Eberly S, deBlieck EA, Oakes D, Lawrence RA. Randomized clinical trial of pacifier use and bottle-feeding or cupfeeding and their effect on breastfeeding. Pediatrics. 2003 Mar;111(3):511-8. doi: 10.1542/peds.111.3.511. PMID 12612229
- [Background] Seema, Patwari AK, Satyanarayana L. Relactation: an effective intervention to promote exclusive breastfeeding. J Trop Pediatr. 1997 Aug;43(4):213-6. doi: 10.1093/tropej/43.4.213. PMID 9283123
- [Background] Lodge CJ, Bowatte G, Matheson MC, Dharmage SC. The Role of Breastfeeding in Childhood Otitis Media. Curr Allergy Asthma Rep. 2016 Sep;16(9):68. doi: 10.1007/s11882-016-0647-0. PMID 27595154
- [Background] Lawrence, R, Lawrence, R (2016) Breastfeeding A Guide for The Medical Professional. Eighth Edition